CLINICAL TRIAL: NCT05417685
Title: Digital Care Programs for Musculoskeletal Health: a Large-scale, Multi-disorder, Observational Study
Brief Title: Digital Care Programs for Musculoskeletal Health
Status: Enrolling by invitation | Type: Observational
Sponsor: Sword Health, SA (Industry)
Responsible Party: Sponsor
Other Study IDs: SH-OBS-MSK-US-01
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Subacute Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Musculoskeletal disorder
  Interventions: Device: Acute and post-acute; Device: Chronic; Device: Post-surgical

INTERVENTIONS:
Device: Acute and post-acute — These programs will cover patients suffering from acute or post-acute musculoskeletal conditions including, but not limited to, shoulder pain (tendinitis/impingement/bursitis), neck pain, low back pain, knee or hip pain/osteoarthritis, which significantly impact their quality of life, to the extent they seek specialised care in direct relation to these disorders.
Device: Chronic — These programs will cover patients suffering from chronic musculoskeletal conditions including, but not limited to, shoulder pain (tendinitis/impingement/bursitis), neck pain, low back pain, knee or hip pain/osteoarthritis, which significantly impact their quality of life, to the extent they seek specialised care in direct relation to these disorders.
Device: Post-surgical — These programs will cover patients submitted to surgery for a given musculoskeletal condition, including, but not limited to, shoulder tendon repair, shoulder replacement, spinal surgery, hip or knee replacement, meniscal repair, knee ligament reconstruction, undergoing physical rehabilitation programs after surgery.

SUMMARY:
The purpose of this study is to create a research repository, composed of data collected in the course of digital care programs for musculoskeletal conditions and musculoskeletal health delivered by SWORD Health to individuals undergoing those programs.

This will allow the investigators to observe the acceptance, engagement and outcomes of programs using this approach in the treatment of multiple musculoskeletal disorders (MSD).

DETAILED DESCRIPTION:
This scientific research was designed to:

* Assess the adoption, engagement and feasibility of digital care programs for musculoskeletal conditions and musculoskeletal health
* Assess the results of digital care programs and compare the costs with the benefits obtained;
* Increase the knowledge on several musculoskeletal conditions, namely how they progress and respond to digital care programs;
* Develop new or improved tools to assist clinicians in the management of these conditions and in helping people achieve better musculoskeletal health

Collection and objective analysis of the collected data will allow:

1. Assess the adoption, engagement and feasibility of digital care programs for musculoskeletal conditions and musculoskeletal health
2. Assess the results of digital care programs and compare the costs with the benefits obtained;
3. Correlate the results with patient's demographic and clinical profiles;
4. Examine the impact of mental health and the behavioral modification components of SWORD Health interventions on disease markers, comorbidities, and productivity;
5. Increase the knowledge on several musculoskeletal conditions, namely how they progress and respond to digital care programs;
6. Develop new or improved tools to assist clinicians in the management of these conditions and in helping people achieve better musculoskeletal health

Clinical outcomes

The primary outcome will be the evolution of patient's clinical condition along the rehabilitation program, objectively estimated through the monitoring data collected using SWORD Phoenix®, as part of patients' supervision routine. Depending on the condition, primary and secondary outcome measures vary.

In any case, this registry will include a complete characterisation of the clinical condition, as well as the periodic assessment of: a) joints' range of motion (collect by the medical device); b) performance indicators (through condition-specific tests); c) patient-reported outcomes (obtained using internationally validated pathology-specific questionnaires); d) pain and fatigue levels (reported by patients by the end of each therapeutic exercise session); e) compliance; f) patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Acute (<12 weeks) or chronic (>12 weeks) musculoskeletal pain involving any of the following body areas: neck, upper and lower back, shoulder, elbow, wrist/hand, hip, knee, ankle OR Recovering from MSK surgery involving the above body areas with indication from their surgeon to engage in a physical therapy program
* Able to understand study procedures and willing to provide informed consent.

Exclusion Criteria:

* Health condition (cardiac, respiratory, neurological, immune) condition incompatible with at least 20 minutes of light to moderate exercise if not cleared by a physician to engage in an exercise program
* Rapidly progressive and new in onset neurological complaints if not cleared by a physician to engage in an exercise program
* Active cancer diagnosis or receiving treatment for cancer if not cleared by a physician to engage in an exercise program
* Significant trauma to the area of pain within the last 12 weeks and functional incapacity and not cleared by a physician to engage in an exercise program
* MSK surgery within the last 12 weeks and not cleared by a physician to engage in an exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: These programs will cover patients suffering from musculoskeletal conditions including, but not limited to, shoulder pain (tendinitis/impingement/bursitis), neck pain, low back pain, knee or hip pain/osteoarthritis, which, irrespective of their duration (acute, post-acute or chronic), significantly impact their quality of life, to the extent they seek specialized care in direct relation to these disorders. The programs will also cover patients submitted to surgery for a given musculoskeletal condition, including, but not limited to, shoulder tendon repair, shoulder replacement, spinal surgery, hip or knee replacement, meniscal repair, knee ligament reconstruction, undergoing physical rehabilitation programs after surgery.
Sampling Method: Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported Pain (NPRS) | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Pain Numerical Rating Scale
Short version of the Disabilities of the Arm, Shoulder and Hand questionnaire | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the short version of the Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH).
  Scoring Formula = ([(sum of n responses)/n] -1)x(25).
Oswestry Disability Index (ODI) | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the Oswestry Disability Index (ODI). \ The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Neck Disability Index (NDI) | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the Neck Disability Index (NDI). For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated as follows: Example:16 (total scored)
  50 (total possible score) x 100 = 32%
Short form of Foot and Ankle Ability Measure (QuickFAAM) | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time, measured through the short form of Foot and Ankle Ability Measure (QuickFAAM). This is a 12-item scale with 5-likert options, the total number of points are added, divided by the total number os possible points and then multiplied by 100.
Short form Hip Osteoarthritis Outcomes Score (HOOS-PS) | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time, measured through the short form Hip Osteoarthritis Outcomes Score (HOOS-PS). This is a 5-item scale with 5-likert options, the total number of points are added, divided by the total number os possible points and then multiplied by 100.
Short form Knee Osteoarthritis Outcomes score (KOOS-PS) | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time, measured through the short form Knee Osteoarthritis Outcomes score (KOOS-PS) This is a 7-item scale with 5-likert options, the total number of points are added, divided by the total number os possible points and then multiplied by 100.
Fear avoidance behaviour | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes of low back pain measured through the Fear Avoidance Beliefs Questionnaire - Physical Activity (FABQ - PA). This is a 5-item scale with 6 likert options. The total number of points are added. Maximum score is 30. Higher scores mean higher fear avoidance (higher scores are worse).
Neck, lower spine, shoulder, elbow, ankle, hip and knee range of motion (ROM) | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through Neck, lower spine, shoulder, elbow, ankle, hip and knee range of motion (ROM) (flexion/extension/abduction/rotation), in degrees, as directly retrieved from the angle measurement tool integrated within the medical device.

SECONDARY OUTCOMES:
Self-reported Pain (VAS) | Baseline and following each exercise session through program completion, an average of 40 sessions
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Visual Analogue Scale for pain
Self-reported fatigue (VAS) | Baseline and following each exercise session until the end of the program
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Visual Analogue Scale for fatigue
Self-reported Surgical intent | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through Numerical rating scale (0-100)
Self-reported consumption of painkillers | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through Self-reported consumption of painkillers (yes/no; Prescription drugs (yes/no); Opioids intake (yes/no)
Anxiety | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through General Anxiety Disorder-7 (GAD-7) is a 7-item scale (scores 0-21)
Depression | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale (0-27)
Work productivity and absenteeism | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through Work Productivity and Activity Impairment Questionnaire (WPAI) assessed by the sub-scores: WPAI overall (combining presenteeism and absenteeism), WPAI work (presenteeism), WPAI time (absenteeism) and WPAI activities (activities of daily living impairment) (scores 0-100%)

OTHER OUTCOMES:
Sessions performed | Measured at the end of the program, an average of 12 weeks
  Number of total exercise sessions performed
Self-reported satisfaction | Baseline, and then at regular intervals (after 9, 18 and 27 sessions) after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  measured through the Net Promoter Score question collected at end of program: "On a scale from 0 to 10, how likely are you to recommend SWORD's programs to a friend or family member?")
Total treatment time | Measured at the end of the program, an average of 12 weeks
  Number of minutes spent on exercise sessions (aggregated)
Average treatment time per week | Measured at the end of the program, an average of 12 weeks
  Average number of minutes spent on exercise per week

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, PhD, Principal Investigator — SWORD HEALTH INC
Locations (1):
- Sword Health, Draper, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and study aggregate results (including anonymised individual patient data) will be made available.
Supporting Information: Study Protocol
Time Frame: The data will become available upon studies publication, for 5 years.
Access Criteria: Study protocol and the aggregate results will be made available as supplementary information or upon reasonable request upon study publication

REFERENCES:
- [Derived] Janela D, Tong X, Pires D, Fonseca H, Costa F. Predicting Pain Outcomes after Digital Care in Chronic Spinal Pain: the roles of Disability, Work Impairment, and Occupation in a Secondary Analysis of a Prospective Clinical Study. Pain Med. 2026 Feb 2:pnag019. doi: 10.1093/pm/pnag019. Online ahead of print. PMID 41629208
- [Derived] C Areias A, G Moulder R, Molinos M, Janela D, Bento V, Moreira C, Yanamadala V, P Cohen S, Dias Correia F, Costa F. Predicting Pain Response to a Remote Musculoskeletal Care Program for Low Back Pain Management: Development of a Prediction Tool. JMIR Med Inform. 2024 Nov 19;12:e64806. doi: 10.2196/64806. PMID 39561359
- [Derived] Areias AC, Janela D, Molinos M, Bento V, Moreira C, Yanamadala V, Cohen SP, Correia FD, Costa F. Exploring the Importance of Race and Gender Concordance Between Patients and Physical Therapists in Digital Rehabilitation for Musculoskeletal Conditions: Observational, Longitudinal Study. J Med Internet Res. 2024 Oct 29;26:e65354. doi: 10.2196/65354. PMID 39470695